CLINICAL TRIAL: NCT06008938
Title: An Observational Post-authorization Long-term Follow-up Study to Characterize the Effectiveness and Safety of HEMGENIX® (Etranacogene Dezaparvovec) in Patients With Hemophilia B
Brief Title: An Observational Cohort Study to Characterize the Effectiveness and Safety of HEMGENIX® in Patients With Hemophilia B
Acronym: IX-TEND 4001
Status: Recruiting | Type: Observational
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Other Study IDs: CSL222_4001; EUPAS106066 (Registry Identifier: EU PAS (ENCePP))
Record Dates: First submitted 2023-08-15; First posted 2023-08-24 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Hemophilia B
Keywords: Hemophilia B; HEMGENIX
MeSH Terms: conditions — Hemophilia B | interventions — Factor IX

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HEMGENIX: Patients with hemophilia B treated with HEMGENIX in countries where HEMGENIX is approved for commercial use.
  Interventions: Genetic: HEMGENIX
- FIX Prophylaxis: Patients with hemophilia B on FIX prophylaxis and enrolled in American Thrombosis and Hemostasis Network (ATHN) Transcends (A Natural History Cohort Study of the Safety, Effectiveness, and Practice of Treatment in People with Non-Neoplastic Hematologic Disorders) Hemophilia Cohort, or a similar registry.
  Interventions: Biological: Factor IX (FIX)

INTERVENTIONS:
Genetic: HEMGENIX — HEMGENIX is a gene therapy medicinal product that aims to deliver a factor IX (FIX) gene expression cassette to the liver of patients with hemophilia B.
  Other Names: Etranacogene dezaparvovec
  Groups: HEMGENIX
Biological: Factor IX (FIX) — FIX prophylaxis therapy
  Groups: FIX Prophylaxis

SUMMARY:
This observational, post-authorization, long-term follow-up study aims to investigate the short and long-term effectiveness and safety of HEMGENIX in patients with hemophilia B. The study will also include a cohort of patients with hemophilia B treated with FIX prophylaxis to enable interpretation of relevant efficacy and safety findings of HEMGENIX.

ELIGIBILITY:
Inclusion Criteria:

* HEMGENIX Cohort:
* - Treatment with commercial HEMGENIX.
* - Have provided signed written informed consent within 3 months before or within 6 months after HEMGENIX treatment, or within 6 months of when the study is initiated at the participating site.
* FIX Prophylaxis Cohort:
* - Adult patients (≥ 18 years) with hemophilia B who have consented and enrolled in ATHN Transcends Hemophilia Cohort (or a similar registry) and are receiving FIX prophylaxis therapy.

Exclusion Criteria:

* HEMGENIX Cohort:
* - The patient population that will be observed in this study must not have been treated with etranacogene dezaparvovec in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hemophilia B who have been treated with HEMGENIX and are enrolled in either the sponsor's study or the ATHN Transcends study NCT04398628 (Hemophilia Cohort, Gene Therapy Outcomes Arm), and patients who receive routine prophylaxis treatment with FIX replacement therapy that are enrolled in the ATHN Transcends study (Hemophilia Cohort, Natural History Arm), or a similar registry. All patients will provide signed informed consent required for participation.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2043-08-01 (Estimated); Study Completion 2043-08-01 (Estimated)

PRIMARY OUTCOMES:
Bleeding Rate (all bleeds) - HEMGENIX Cohort | During the 52 weeks following stable FIX expression (6 to 18 months) in the follow-up period and at Months 6 to: 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, and 180 after HEMGENIX treatment.
  Annualised Bleeding Rate (ABR) for all bleeds

SECONDARY OUTCOMES:
Bleeding Rate (specified bleed types) - HEMGENIX Cohort | During follow-up period (52 weeks following stable FIX expression [6 to 18 months]), and at Months 6 to: 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, and 180 after HEMGENIX treatment.
  ABR for spontaneous, FIX-treated, traumatic, and joint bleeds
Zero bleeds - HEMGENIX Cohort | During follow-up after HEMGENIX treatment, up to 180 months
  Number of patients with zero bleeds
Correlation analysis - HEMGENIX Cohort | Over the 6 to: 18, 24, 36, 48, 60, 72, 96, 108, 120, 132, 144, 156, 168, and 180 months after HEMGENIX treatment.
  Correlation analysis of ABR as a function of mean FIX activity.
Bleeding Rate - FIX Prophylaxis Cohort | In the period Months 0 to: 12, 18, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, and 180 Months.
  ABR (total, spontaneous, FIX-treated, traumatic, and joint bleeds)
FIX activity - HEMGENIX Cohort | Day 1, Week 6, and Months 6, 12, 18, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, and 180 after HEMGENIX treatment.
  Mean uncontaminated endogenous FIX activity (%)
Annualized consumption of FIX replacement therapy - HEMGENIX Cohort | During the follow-up periods (52 weeks following stable FIX expression [6 to 18 months], & at Months 0 to: 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, and 180), & at yearly intervals (ie, at 0 to 1 yr, 1 to 2 yrs, etc, up to 14 to 15 yrs).
  Mean annualized consumption (IU/kg/Yr) of FIX replacement therapy (including FIX replacement for various clinical scenarios eg, prophylaxis, spontaneous bleeding events, medical procedures, surgery, and trauma).
Annualized consumption of FIX replacement therapy - FIX Prophylaxis Cohort | At Months 0 to: 12, 18, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, and 180.
  Mean annualized consumption (IU/kg/Yr) of FIX replacement therapy (including FIX replacement for various clinical scenarios eg, prophylaxis, spontaneous bleeding events, medical procedures, surgery, and trauma).
Number of patients remaining free of previous continuous routine prophylaxis - HEMGENIX Cohort | At Months 6 to: 18, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, and 180 after HEMGENIX treatment.
  Number and proportion of patients remaining free of previous continuous routine prophylaxis (FIX replacement therapy)
Target joints occurrence - HEMGENIX Cohort | After HEMGENIX treatment, during the follow-up periods (52 weeks following stable FIX expression [6 to 18 months], and at Months 6 to: 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, and 180).
  The annualized occurrence of target joints (defined as 3 or more spontaneous bleeding events into a single joint within a consecutive 6-month period).
Target joints resolution - HEMGENIX Cohort | During the follow-up period, up to 180 months
  The percentage of resolution of target joints (target resolution is defined as a recorded target joint with 2 or fewer spontaneous bleeding events within a consecutive 12-month period).
Target joints - FIX Prophylaxis Cohort | From Months 0 to 12, 18, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, and 180.
  The annualized occurrence of target joints
Related Serious Adverse Events (SAEs) - number | During 15 years of follow-up
  Incidence (number) of related SAEs
Related SAEs - percent | During 15 years of follow-up
  Incidence (percent) of related SAEs
Adverse Events of Special Interest (AESIs) - number | During 15 years of follow-up
  Incidence (number) of AESIs
AESIs - percent | During 15 years of follow-up
  Incidence (percent) of AESIs

CONTACTS AND LOCATIONS:
Overall Officials: Global Program Director, Study Director — CSL Behring
Locations (10):
- American Thrombosis and Hemostasis Network, Rochester, New York, United States
- Medical University Vienna, Vienna, Austria
- Aarhus Universitetshospital, Århus N, Denmark
- France (3):
  - Centre Hospitalier Universitaire de Brest / CHU Morvan, Brest
  - Centre Régional de Traitement de l'Hémophilie, Nantes
  - CHU Nancy - Hôpital Brabois, Vandœuvre-lès-Nancy
- Germany (2):
  - Klinik für Angiologie/ Hämostaseologie, Berlin
  - Hannover Medical School, Hanover
- Hospital Alvaro Cunqueiro Dr. Manuel Rodriquez-Lopez, Vigo, Spain
- University Hospital Bern Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider requests to share Individual Patient Data (IPD) from systematic review groups or bona-fide researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.
Supporting Information: Study Protocol, SAP
Time Frame: IPD requests may be submitted to CSL no earlier than 12 months after publication of the results of this study via an article made available on a public website.
Access Criteria: Requests may only be made by systematic review groups or bona-fide researchers whose proposed use of the IPD is non-commercial in nature and has been approved by an internal review committee.
  An IPD request will not be considered by CSL unless the proposed research question seeks to answer a significant and unknown medical science or patient care question as determined by CSL's internal review committee.
  The requesting party must execute an appropriate data sharing agreement before IPD will be made available.